CLINICAL TRIAL: NCT06172946
Title: Effect of Inspiratory Muscle Training Versus Transcutaneous Electrical Diaphragmatic Stimulation on The Severity of Copd
Brief Title: Effect of Powerbreath Versus Transcutaneous Electrical Diaphragmatic Stimulation on The Severity of Copd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed El-Moatasem Mohamed, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004626
Record Dates: First submitted 2023-12-03; First posted 2023-12-15 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- INSPIRATORY MUSCLE TRAINING (Experimental): Power Breathe:
  (3times/week for 8 weeks) The patient should inhale and exhale through the mouthpiece 30 times maximum. The training load is adjustable and should be set at a level appropriate for the patient to effectively train the inspiratory muscles. (Lázaro et al., 2021)
  Interventions: Device: powerbreath
- TRANSCUTANEOUS ELECTRICAL DIAPHRAGMATIC STIMULATION (Active Comparator): Transcutaneous electrical Diaphragmatic Stimulation(TEDS):
  (3times/week for 8 weeks) During each session, rectangular electrodes were placed on the parasternal region beside the xiphoid process; the sixth and seventh intercostal spaces in line with the mid-axillary line. The electrical current is pulsed, biphasic and symmetric, with the following parameters: frequency of 30 Hertz; 0.4ms phase width, rise time of 0.7 seconds; respiratory rate of 14 rpm; intensity is the minimum necessary to obtain diaphragm muscle contraction. TEDS intensity was gradually increased until visible muscle contraction was observed. (Hsin et al., 2022)
  Interventions: Device: TRANSCUTANEOUS ELECTRICAL DIAPHRAGMATIC STIMULATION

INTERVENTIONS:
Device: powerbreath — Previous studies have confirmed the efficacy of implementing IMT as part of a RR program in a certain profile of patients with COPD, showing improvements in maximum inspiratory pressure, perception of well-being, and other respiratory diseases, and dyspnea during exercise. (Gandullo et al., 2022)
  Arms: INSPIRATORY MUSCLE TRAINING
Device: TRANSCUTANEOUS ELECTRICAL DIAPHRAGMATIC STIMULATION — Transcutaneous electrical diaphragmatic stimulation (TEDS) has been used to improve respiratory muscle strength in patients with respiratory muscle weakness. A previous study reported that patients with chronic obstructive pulmonary disease (COPD) showed increased lung volume and oxygen saturation after a single session of TEDS. (Hsin et al., 2022)
  Arms: TRANSCUTANEOUS ELECTRICAL DIAPHRAGMATIC STIMULATION

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common and treatable disease characterized by progressive airflow limitation and tissue destruction. It is associated with structural lung changes due to chronic inflammation from prolonged exposure to noxious particles or gases most commonly cigarette smoke.

POWERbreathe device (POWER-breathe International Ltd., Southam, Warwickshire, UK) is an inspiratory muscle training and this device has recently shown benefits on pulmonary function. Also, the POWER-breathe® device's effects on the strength of the diaphragm muscle and minimize muscle weakness and wasting in COPD patients.

Neuromuscular electrical stimulation (NMES) is commonly used in physical therapy to increase muscle strength and promote muscle hypertrophy. NMES applied to respiratory rehabilitation is called transcutaneous electrical diaphragmatic stimulation (TEDS).

DETAILED DESCRIPTION:
sixty Patients will be assigned randomly into two equal groups with pre and post treatment protocol application.

Group A:

Thirty patients will be treated by power breathe along with their prescribed medication.

Group B:

Thirty patients will be treated by Transcutaneous electrical Diaphragmatic Stimulation (TEDS) along with their prescribed medication.

ELIGIBILITY:
Inclusion Criteria:

* The patient selection will be according to the following criteria:

  1. Male patients diagnosed with stage 2&3 COPD.
  2. All patients are under full medical control.
  3. Their ages will range from forty-five to sixty-five years.
  4. Patients with BMI from 25-29.9 kg/m2

Exclusion Criteria:

* Patients with the following criteria will be excluded from the study:

  1. Lack of language or cognitive abilities to fill out questionnaire.
  2. Patients with cardiac pacemaker.
  3. Contraindications for inspiratory muscle training (e.g. a history of recent lung surgery, recent pulmonary embolism, history of recurrent spontaneous pneumothorax, other serious lung disease).
  4. Existing arterial aneurysm.
  5. Clinical signs of unstable cardiac event (eg. congestive heart failure).
  6. Patients with malignant disease.
  7. Acute COPD exacerbation within the last 4 weeks.
  8. Any need for supplemental oxygen.
  9. Patients with Gastro-esophageal reflux disease.
  10. Patients with active Hemoptysis.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
The COPD Assessment Test (CAT) | COPD Assessment Test will be measured at baseline, and it will be measured again after eight weeks
  The COPD Assessment Test(CAT) is validated questionnaire consisting of eight items, which evaluate the most burdensome symptoms and limitations of the patients. The score for each item ranges from 0 to 5 and the total score (0-40)

SECONDARY OUTCOMES:
Pulmonary function: By Spirometry Device: | Pulmonary function: By Spirometry Device: forced vital capacity will be measured at baseline, and it will be measured again after eight weeks
  • Pulmonary function: By Spirometry Device: it measure ventilatory functions. forced vital capacity (FVC)
Pulmonary function: By Spirometry Device: | Pulmonary function: By Spirometry Device: forced expiratory volume in one second will be measured at baseline, and it will be measured again after eight weeks
  • Pulmonary function: By Spirometry Device: it measure ventilatory functions. forced expiratory volume in one second (FEV1)
Pulmonary function: By Spirometry Device: | Pulmonary function: By Spirometry Device: forced expiratory volume in one second/forced expiratory volume will be measured at baseline, and it will be measured again after eight weeks
  • Pulmonary function: By Spirometry Device: it measure ventilatory functions. forced expiratory volume in one second/forced expiratory volume (FEV1/FVC)
Pulmonary function: By Spirometry Device: | Pulmonary function: By Spirometry Device: forced expiratory flow will be measured at baseline, and it will be measured again after eight weeks
  • Pulmonary function: By Spirometry Device: it measure ventilatory functions. forced expiratory floe(FEF25-75%)
Diaphragmatic Thickness: By Ultrasonography: | Diaphragmatic Thickness: By Ultrasonography:will be measured at baseline, and it will be measured again after eight weeks
  • Diaphragmatic Thickness: By Ultrasonography: provides a simple and non-invasive means of assessing diaphragmatic function. (Boussuges et al., 2020)
Measuring functional capacity: By Six-minute walk test (6MWT): | Measuring functional capacity: By Six-minute walk test (6MWT)::will be measured at baseline, and it will be measured again after eight weeks
  • Measuring functional capacity: By Six-minute walk test (6MWT): is a self paced submaximal field exercise test , It will be performed according to the standard procedure is administered in a 30 meter hallway. (Launois et al., 2012 and ATS statement2002)
Modified Medical Research Council dyspnea scale (mMRC dyspnea scale): | Modified Medical Research Council dyspnea scale (mMRC dyspnea scale):will be measured at baseline, and it will be measured again after eight weeks
  • Dyspnea: By Modified Medical Research Council dyspnea scale (mMRC dyspnea scale): It is a 5 point scale based on degrees of variable physical activities that precipitate dyspnea with a score ranging from 0 to 4. (Richards, 2017)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt